CLINICAL TRIAL: NCT07049757
Title: Healthy Family Project: Ending Tobacco Use and Smoke Exposure in Asian American Communities
Brief Title: Healthy Family Project: Tobacco Use and Smoke Exposure in Asian American Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 24634; NCI-2025-00206 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Tobacco-Related Carcinoma; Smoking Cessation
Keywords: Third-hand Smoke
MeSH Terms: conditions — Smoking Cessation | interventions — Educational Status; Methods; Surveys and Questionnaires; Urine Specimen Collection; Interviews as Topic; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Development (Focus group + Interview) (Experimental): To achieve information gathering and preliminary adaptation design to prepare for the randomized clinical trial, focus groups and individual interviews with 24 participants (6 Chinese current smokers; 6 former smokers who have stopped smoking within the past 2 years; and 12 family/household members living with a current/former smoker) to review the newly developed or updated intervention materials. The Community Advisory Board (CAB) will also be involved in providing input.
  Interventions: Other: Focus Group
- Arm I: Quit Smoking for a Healthy Family Group (QS) (Active Comparator): Participants attend two QS educational sessions over 45-60 minutes one month apart and receive two follow-up phone calls over 15-30 minutes 1-2 weeks after each session over 6 weeks. Participants also receive a Healthy Family Action Plan as well as a smoking cessation resource guide and set goals on study. Participants then receive THS education and cleaning strategies at 6 months after the initial QS curriculum. Additionally, participants undergo urine sample collection throughout the study and non-smoking family/household members will wear a silicone wristband for 2 days at each assessment.
  Interventions: Other: Smoking cessation education; Behavioral: Survey Administration; Behavioral: Telephone-Based Intervention; Procedure: Urine Specimen Collection; Other: Silicone Wrist Band; Other: Interview
- Arm II: Smokefree Family Living Group (SFL) (Experimental): Participants attend two QS educational sessions over 45-60 minutes one month apart and receive two follow-up phone calls over 15-30 minutes 1-2 weeks after each session over 6 weeks. During the second QS educational session, participants receive THS education and cleaning strategies. Participants also receive a Healthy Family Action Plan as well as a smoking cessation resource guide and set goals on study. Additionally, participants undergo urine sample collection throughout the study and non-smoking family/household members will wear a silicone wristband for 2 days at each assessment.
  Interventions: Other: Smoking cessation education; Behavioral: Survey Administration; Behavioral: Telephone-Based Intervention; Procedure: Urine Specimen Collection; Other: Silicone Wrist Band; Other: Interview

INTERVENTIONS:
Other: Smoking cessation education — Quit Smoking for a Healthy Family (QS) and Smokefree Family Living (SFL) education sessions to promote smoking cessation and reduce tobacco smoke exposure.
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Behavioral: Survey Administration — Administered for ancillary studies
  Other Names: Questionnaires
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Behavioral: Telephone-Based Intervention — Participants will receive follow-up calls
  Other Names: Telephone-Based Follow-up
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Procedure: Urine Specimen Collection — Undergo urine sample collection at baseline
  Other Names: Urine Sample
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Other: Silicone Wrist Band — Non-smoking family/household members will wear a silicone wristband for 2 days at each assessment for ancillary studies
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Other: Interview — Selected participants will take part in an interview for ancillary studies
  Other Names: In-depth interview
  Arms: Arm I: Quit Smoking for a Healthy Family Group (QS); Arm II: Smokefree Family Living Group (SFL)
Other: Focus Group — Participants will review and comment on materials under development to be used in randomized clinical trial.
  Arms: Intervention Development (Focus group + Interview)

SUMMARY:
This study evaluates whether the Smokefree Family Living (SFL) intervention improves quit rates (smoking cessation) and exposure to tobacco contamination that stays in items such as, carpets, walls, and furniture, even after the smoke has cleared (third-hand smoke (THS)) among Chinese American smokers and their non-smoking household members. Smoking remains high among Chinese American males with limited ability to speak English. This causes the non-smoking household members to be exposed to THS, which contains many of the same harmful components as smoking and becomes more toxic as it ages. SFL is tailored for Chinese Americans and combines the contents of the Quit Smoking for a Healthy Family (QS) intervention with additional THS education and cleaning strategies. QS focuses on smoking cessation through educational sessions and support. THS education and cleaning strategies provide information on THS and how to clean the home for THS. SFL may help Chinese American smokers and their non-smoking household members learn about the importance of quitting and the dangers of THS, this may improve smoking cessation and reduce THS exposure

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Integrate the original "Quit Smoking for a Healthy Family" (QS) curriculum with the third-hand smoke education and cleaning intervention (THS) into a new intervention titled "Smokefree Family Living" (SFL) for Chinese immigrant families and household members.

II. Examine the efficacy of SFL by measuring smoking cessation rates at six months and the reduction in third-hand smoke exposure among smokers and nonsmoking household member participants, respectively, using a 2-arm randomized trial targeting 320 smoker-household member dyads from the Chinese American communities.

SECONDARY OBJECTIVE:

I. Examine individual and social pathways mediating the outcomes for cessation attempts, abstinence, and tobacco smoke exposure.

EXPLORATORY OBJECTIVES:

I. Explore the long-term impacts of the THS education and the timing of the accessibility of the THS intervention by examining time to first 30-day quit attempts and duration of quit attempts after exposure to THS intervention in both intervention groups of a subsample available for 12-month follow-up.

II. To compare the long-term efficacy of the SFL and QS interventions in sustaining smoking cessation and reducing tobacco smoke exposure.

III. To evaluate the feasibility and effectiveness of using silicone wristbands to measure third-hand smoke (THS) exposure among non-smoking household members of Chinese American smokers participating in the study.

IV. Assess the behavioral changes related to smoking and smoke exposure, as well as the psychosocial impact of the interventions on participants and their household members.

OUTLINE:

A family-based intervention development phase prior to the randomized study will integrate the original "Quit Smoking for a Healthy Family" (QS) curriculum of the Healthy Family Project with the third-hand smoke education and cleaning intervention (THS) into a newly integrated intervention named "Smokefree Family Living" (SFL) for Chinese immigrant families and household members. Information collected from this group will be used to refine and develop the final SFL intervention used in the subsequent clinical trial. These participants will not be included in final study analyses.

Participants enrolled after the focus group data has been evaluated for implementation will be randomized to 1 of 2 arms.

ARM I: Participants attend two QS educational sessions over 45-60 minutes one month apart and receive two follow-up phone calls over 15-30 minutes 1-2 weeks after each session over 6 weeks. Participants also receive a Healthy Family Action Plan as well as a smoking cessation resource guide and set goals on study. Participants then receive THS education and cleaning strategies at 6 months. Additionally, participants undergo urine sample collection throughout the study.

ARM II: Participants attend two QS educational sessions over 45-60 minutes one month apart and receive two follow-up phone calls over 15-30 minutes 1-2 weeks after each session over 6 weeks. During the second QS educational session, participants receive THS education and cleaning strategies. Participants also receive a Healthy Family Action Plan as well as a smoking cessation resource guide and set goals on study. Additionally, participants undergo urine sample collection throughout the study.

After completion of study intervention, participants are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

All Participants (Lay Health Workers, Smokers, Family Participants, and Post-Trial Household Member Group Interview Participants):

1. Must be 18 years of age or older.
2. Must self-identify as Chinese or of Chinese descent (ethnic or cultural identification, not national origin).
3. Must be able to understand in spoken Chinese (Cantonese and/or Mandarin) or English.
4. Able to attend educational sessions in person or via video conferencing.
5. Ability to understand and the willingness to sign a written informed consent document.

Lay Health Workers:

1. Must have experience or interest in community outreach and education.
2. Must demonstrate proficiency in language (Cantonese and/or Mandarin or English) sufficient to deliver study materials and interact with participants.
3. Must be affiliated with the Chinese Community Health Resource Center (CCHRC) or recruited through community networks.
4. Must agree to participate in training and intervention delivery activities as outlined in the study protocol.

Smokers (Participants who are current smokers):

1. Must have smoked within the past 30 days, either daily or occasionally.
2. Must have a non-smoking household member.

Family Participants (Non-smoking family/household members):

1. Must live in the same household as the smoker participant.
2. Must not have used any tobacco products in the past 30 days.

Post-Trial Household Member Group Interview Participants:

1. Living in the same household with the smoker-household member dyad participant being interviewed or considered as a household member.

Exclusion Criteria:

Lay Health Workers, Smokers (Participants who are current smokers) and Family Participants (Non-smoking Family/household members):

1. Currently participating in another smoking cessation program.
2. Non-residents of California.
3. Participants unwilling to provide follow-up contact for assessments at 6 and 12 months.

Lay Health Workers:

1. Lack of willingness or ability to complete training or deliver intervention sessions as required by the study protocol.
2. Inability to maintain confidentiality and professionalism during interactions with study participants.
3. Active participation in conflicting research studies or programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who have quit smoking at 6 months | 6 months
  The smoking cessation rate is defined as the proportion of smokers who report quitting smoking, with biochemically verified 30-day point prevalent abstinence at the 6-month follow-up. Smoking rates will be reported by arm.

SECONDARY OUTCOMES:
Change in levels of tobacco smoke biomarkers for second-(SHS)hand smoke exposure | Up to 6 months
  The change in level of tobacco smoke exposure will be assessed among non-smoking family/household members by reviewing levels of urinary 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) at baseline and at 6 months.
Proportion of participants who have quit smoking at 12 months | Up to 12 months
  The smoking cessation rate is defined as the proportion of smokers who report quitting smoking, with verified 30-day point prevalent abstinence by biochemical markers (e.g., urinary NNAL and cotinine tests) at the 12-month follow-up. Smoking rates will be reported by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No